CLINICAL TRIAL: NCT05598580
Title: Functional Cure Strategy and Clinical Study of AIDS--Study on the Reduction of HIV Viral Reservoir by Immunomodulators (IMs)
Brief Title: Immunomodulators on HIV-1 Reservoir
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022IMs
Record Dates: First submitted 2022-10-26; First posted 2022-10-28 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Lenalidomide (Experimental): Lenalidomide capsules (25 mg) were administered orally on days 1-21 of a 28-day cycle for 24 weeks with continuous antiretroviral therapy. After that, participants will be monitored for another 24 weeks.
  Interventions: Drug: Lenalidomide
- Adenosylmethionine (Experimental): Adenosylmethionine capsules (1000 mg, twice a day) were administered orally for 24 weeks with continuous antiretroviral therapy. After that, participants will be monitored for another 24 weeks.
  Interventions: Drug: Adenosylmethionine
- Control (No Intervention): Participants will continue to receive antiretroviral therapy without other intervention and be monitored for 48 weeks.

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide capsules (25 mg) were administered orally on days 1-21 of a 28-day cycle for 24 weeks with continuous antiretroviral therapy.
  Arms: Lenalidomide
Drug: Adenosylmethionine — Adenosylmethionine capsules (1000 mg, twice a day) were administered orally for 24 weeks with continuous antiretroviral therapy.
  Arms: Adenosylmethionine

SUMMARY:
The goal of this clinical trial is to learn about the function of immunomodulators in reducing HIV reservoir. The main questions it aims to answer are:

* Are immunomodulators able to reduce HIV reservoirs?
* How do immunomodulators reduce HIV reservoirs? Participants will be randomly and equally divided into three groups, one control group and two trial groups. All three groups will continue to receive antiretroviral therapy. The two experimental groups will additionally be given different immunomodulators lenalidomide and adenosylmethionine, respectively. The effectiveness of immunomodulatory agents in reducing viral reservoirs will be explored by comparing relevant indicators in the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age ≥ 18 and ≤ 65 years.
* HIV-1 infection, confirmed by any licensed rapid HIV test and then a licensed Western blot.
* Virologic suppression defined as HIV-1 RNA level below the limit of quantification prior to study entry.
* CD4+ T cell count > 200 cells/mm3 prior to study entry.
* Ability and willingness of participant or legal representative to provide written informed consent and attend study visits as scheduled at a participating site. Willingness of participant to accept the side effects of drugs.
* All participants of reproductive potential, who are participating in sexual activity that could lead to pregnancy, must agree to use at least one reliable method of contraception from 4 weeks before the start of the study to 4 weeks after the end of the study.

Exclusion Criteria:

* Breastfeeding or pregnancy, or planned pregnancy during the study.
* Poor treatment adherence.
* Use of immunomodulators or systemic cytotoxic chemotherapy ≤ 6 months prior to study entry.
* Any current diagnosis or past history of a significant cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, neuropsychiatric, psychiatric, or other serious illness. The following laboratory values obtained prior to entry:

  * Absolute neutrophil count (ANC) ≤ 1000/mm3
  * Platelets ≤ 75,000/mm3
* Known allergy/sensitivity or any hypersensitivity to components of study drug or their formulation.
* Unwilling to provide written informed consent.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
HIV reservoirs | 48 weeks
  The size of the HIV reservoir in blood determined by HIV-DNA and CA-HIV-RNA.
Decreased inflammatory factors in HIV-infected patients | 48 weeks
  The following inflammatory cytokines: interferon-alpha (IFN-α), TNF-α, IL-1, IL-6.

SECONDARY OUTCOMES:
T-cell subsets | 48 weeks
  Absolute CD4+ and CD8+ T-cell counts and CD4/CD8 ratio were measured on peripheral blood mononuclear cells.
Immune activation | 48 weeks
  Immune activation measured by the percentage of human leukocyte antigen-DR isotype (HLA-DR) and CD38 expressing T-cells in blood.
Gut microbiome | 48 weeks
  Diversity and composition of gut microbiome.
Tolerability and safety outcomes | 48 weeks
  Discontinuation and occurrence of adverse event.

CONTACTS AND LOCATIONS:
Overall Officials: Biao Zhu, Principal Investigator — Zhejiang University
Locations (1):
- the first affiliated hospital of Zhejiang university school of medicine, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No